CLINICAL TRIAL: NCT06410781
Title: Effect of Radial Extracorporeal Shockwave Therapy on Ultrasonography Changes in Patients With Iliotibial Band Syndrome
Acronym: ITB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nabil Mahmoud Ismail Abdel-Aal, principle investigator nabil mahmoud ismail abdel-aal, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004959
Record Dates: First submitted 2024-05-08; First posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Iliotibial Band Syndrome
Keywords: iliotibial band syndrome; Radial Extracorporeal Shockwave; ultrasonography changes
MeSH Terms: conditions — Iliotibial Band Syndrome

STUDY DESIGN:
Intervention Model Description: Radial Extracorporeal Shockwave Therapy and traditional therapy
Who Masked: Investigator, Outcomes Assessor
Masking Description: opaque sealed envelope
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radial Extracorporeal Shockwave (Experimental): thirty patients with iliotibial band syndrome will receive Radial Extracorporeal Shockwave and traditional therapy three times a week for six weeks.
  Interventions: Other: Radial Extracorporeal Shockwave; Other: traditional therapy
- traditional therapy (Active Comparator): Thirty patients with iliotibial band syndrome will receive traditional therapy three times a week for six weeks.
  Interventions: Other: traditional therapy

INTERVENTIONS:
Other: Radial Extracorporeal Shockwave — Treatment procedure will be initiated by palpation to locate the painful area around the lateral femoral condyle and the lateral side of the thigh. The therapist uses the principle of clinical focusing where the patient guides the therapist to the most painful area. The area will be treated in a circumferential pattern, starting at the point of maximum pain. At each of the session a total of 4600 pulses will be applied. RESWT will start with 500 pulses at (2 Bar) with the frequency of 15 Hz to the lateral femoral condyle to adjust to treatment.An additional 2000 pulses will be applied at (2- 4 Bar), 15 Hz, depending on pain tolerance. in addition,stretching exercise, manual therapy, and ultrasound on the iliotibial band.
  Arms: Radial Extracorporeal Shockwave
Other: traditional therapy — the patients will receive traditional therapy in the form of stretching exercise, manual therapy and ultrasound on iliotibial band.

SUMMARY:
this study will be conducted to investigate the effects of radial extracorporeal shockwave therapy on ultrasonography changes, pain intensity, pain pressure threshold and lower limb function in patient with iliotibial band syndrome

DETAILED DESCRIPTION:
Iliotibial Band Syndrome is an overuse injury that affect the lateral aspect of the knee. It is common in endurance sport activities such as running and cycling. It is the most common running injury of the lateral knee. ITBS is a non-traumatic overuse injury caused by friction/rubbing of the distal portion of the iliotibial band (ITB) over the lateral femoral epicondyle with repeated flexion and extension of the knee. Females are twice as likely to sustain ITBS compared to male due to sex differences in frontal and transverse plane hip and knee joint angles.An alternative treatment strategy of ITBS is radial extracorporeal shockwave therapy (RESWT). It is considered safe as it results in minor adverse effects including worsening of symptoms over a short period, reversible local swelling, redness and hematoma. RESWT has also shown to be effective in the treatment of several chronic musculoskeletal pain conditions such as lateral epicondylitis, Achilles tendinopathy, plantar fasciitis, patellar tendinopathy, calcific tendinitis of the shoulder and chronic proximal hamstring tendinopathy. sixty patients with iliotibial band syndrome will be assigned randomly to two groups; the first one will receive radial extracorporeal shockwave and traditional therapy, the second one will receive traditional therapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Sixty patients suffer from ITBS.
* The age of patients ranges from (18-55) years.

Exclusion Criteria:

* Signs or symptoms of other pathologies of the knee.
* Previous treatment for ITBS in the last 6 months.
* Use of NSAID's or analgesics later than two weeks before baseline.
* Previous surgery on the affected knee.
* Pregnancy.
* Rheumatic disease.
* Previous shockwave treatment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-20 (Estimated); Primary Completion 2024-11-20 (Estimated); Study Completion 2024-11-20 (Estimated)

PRIMARY OUTCOMES:
iliotibial band thickness | up to six weeks
  ultrasonography device will be used to assess iliotibial band thickness

SECONDARY OUTCOMES:
pain intensity | up to six weeks
  The visual analog scale (VAS) will be used to assess pain intensity. Scores are based on self-reported measures of symptoms that are recorded with a single handwritten mark placed at one point along the length of a 100mm line that represents a continuum between the two ends of the scale "no pain" on the left end of the scale and the "worst pain" on the right end of the scale.
pressure pain threshold | up to six weeks
  pressure algometer will be used to assess pressure pain threshold
lower extremity function | up to six weeks
  The lower extremity functional scale is a well-known and validated patient-rated outcome measure that can be used to measure lower extremity function. The score consists of 20 questions, which are subdivided into 4 groups. These groups consist of activities with increasing physical demands. Questions on activity vary from walking between rooms to running on uneven ground. Each item is scored on a scale of 0 to 4, with a higher score indicating better function. The total score ranges from 0 to 80, with higher scores indicating better lower limb function